## Official title of the study:

## Factors Associated with Pain Level Experience During Orthodontic Treatment

NCT Number: Not Available

Date of the document: 04 February 2021

## Inform Consent for the Investigation

From UAX Innovation and Advanced Specialty Dental Clinic

## Research Title: Research Title

Principle Investigator: Dra. CHIA JUNG, LEE

Introduction - This research will focus on how the patient experience the level of pain during orthodontic treatment and how they managed the pain.

**Purpose of Research** - The purpose of this research is to find if there is a correlation of the pain level in patient with different gender, age, orthodontic treatment type and oral hygiene level. This will help us understand in general how did the patient cope with orthodontic treatment and facilitate the explanation of pain experiences in general to patients who are expected to be treated orthodontically.

**Duration** - The survey should take about 5 to 7 minutes to complete.

Participation - If you agree to participate, a researcher will send you a link to complete the survey. The survey asks your opinions about your pain level experiences during orthodontic treatment and basic information (for example, gender, age, duration and type of orthodontic treatment, oral hygiene routine). The survey will be completed during your orthodontic treatment.

Confidentiality - The data provided by the participant will be considered strictly confidential and will not be given to others without written permission from the participant. Your name will never be used in any reports of this research. What you tell us will be used for final reports, articles in magazines and professional journals, and public talks. The results from this study may be used by researchers in future projects. Please let the researchers know if you would like a report of what we learn.

**Right to Refuse or Discontinue** - The participant has the right to discontinue or decline the participation in the research anytime he/she feels to do so.

Your confidentiality will be respected. However, research records identifying you may be inspected in the presence of the Investigator to their tutors. No information or records that disclose your identity will be published without your consent, nor will any information or records that disclose your identity be removed or released without your consent unless required by law. Even if you decide to stop participating, the information you have provided will be kept and may be used in this study, unless you specifically request otherwise.

**Questions about this study** - If you have any questions about the study, or any concerns or complaints about your rights as a research participant and/or your experiences while participating in this study, please contact: <a href="mailto:clee@myuax.com">clee@myuax.com</a>

YOU WILL HAVE AN OPPORTUNITY JOING A RAFFLE TO WIN AN ORTHODONTIC CLEANING KIT TO THANK YOU FOR THE PARTICIPATION!



ALFONSO X EL SABIO UNIVERSITY Innovation and Advanced Specialty Clinic Orthodontic Department

clee@myuax.com (34) 914 402 330